CLINICAL TRIAL: NCT01863199
Title: A Clinical Trial to Assess the Impact of Home Monitoring to Decrease the Treatment Burden for Neovascular Macular Degeneration (the LIBERTY Study).
Brief Title: Impact of Home Monitoring to Decrease the Treatment Burden for Neovascular Age-related Macular Degeneration (AMD)
Acronym: Liberty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Retinal Consultants of Arizona (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28727
Record Dates: First submitted 2013-05-20; First posted 2013-05-27 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: Wet AMD; AMD; Choroidal neovascularization; Neovascular membrane
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Ranibizumab; Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lucentis every 4 weeks (Active Comparator): Lucentis 0.5mg administered intravitreally every four weeks for 12 months
  Interventions: Drug: Lucentis every 4 weeks
- Lucentis every 12 weeks (Active Comparator): Lucentis 0.5mg administered intravitreally every 12 weeks
  Interventions: Drug: Lucentis every 12 weeks
- Treat and extend (Experimental): Lucentis 0.5mg will be administered on an as needed basis after a loading dose using a treatment extending protocol and home monitoring.
  Interventions: Drug: Lucentis (Treat and extend)

INTERVENTIONS:
Drug: Lucentis (Treat and extend) — Lucentis 0.5mg will be administered on an as needed basis after a loading dose using a treatment extending protocol and home monitoring.
  Arms: Treat and extend
Drug: Lucentis every 4 weeks — Lucentis 0.5mg administered intravitreally every four weeks for 12 months
  Arms: Lucentis every 4 weeks
Drug: Lucentis every 12 weeks — Lucentis 0.5mg administered intravitreally every twelve weeks for 12 months
  Arms: Lucentis every 12 weeks

SUMMARY:
A study to use in home technology to reduce the burden of in office visits and injections.

DETAILED DESCRIPTION:
Without frequent measurement of vision to monitor disease progression some people may be under-treated, while others over-treated. Under-treatment can lead to severe and irreversible disease progression and associated loss of vision. Over-treatment is expensive, uncomfortable and potentially increases the risk of complications. A self-monitoring device such as DigiSight can help subjects keep close control of their treatment, but alleviate the burden of in office monitoring visits. A decreased number of office visits in combination with the home self-monitoring may provide an effective alternative dosing regimen, allowing the physician and subject to closely track the disease progression and treatment effect without the demands of monthly or frequent visits to the office.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Choroidal neovascular membrane (CNV) secondary to AMD, as confirmed by the patient's medical history and a documented diagnosis of CNV
* The study eye must have received at least 3 anti-Vascular endothelial growth factor (VEGF) treatments prior to the screening visit, with at least 2 anti-VEGF treatments over the preceding 3 months.
* Best-corrected visual acuity (BCVA) of 20/32 to 20/200 Snellen equivalent in the study eye
* Noted presence of intra- or sub-retinal fluid on OCT in the study eye
* Adequate pupillary dilation to permit thorough ocular examination and testing in both eyes
* Proficiency in using the DigiSight SightBook™ mobile vision assessment tool on study-supplied Apple iPad or iPod device

Exclusion Criteria:

* CNV in the study eye due to any reason other than AMD
* Active uncontrolled glaucoma
* Had any intraocular surgeries in the study eye within 3 months of enrollment or are known or likely candidates for intraocular surgery (including cataract surgery) in the study eye within 1 year of enrollment
* Acute or chronic ocular or periocular infection in the study eye, uveitis or ocular inflammation in the study eye
* Received Photo Dynamic Therapy (PDT) in the study eye within 60 days, or laser photocoagulation within 14 days prior to screening
* Currently using any periocular or intravitreal steroids within 3 months prior to screening (study eye)
* Unstable or severe cardiovascular disease, e.g., congestive heart failure (New York Heart Association Functional class III/IV), myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina, or critical limb ischemia
* Poorly controlled diabetes
* Cerebrovascular disease within 12 months prior to Screening
* Dementia or neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease)
* Received any investigational product within 30 days prior to Screening
* Inability to properly use the SightBook™ app

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 12 months
  Best corrected visual acuity (BCVA), as assessed by the number of letters read correctly on the Early Treatment Diabetic Retinoptahy Study (ETDRS) eye chart at a starting test distance of 4 meters, at Months 3, 6, 9 and 12

SECONDARY OUTCOMES:
Central foveal thickness | 12 months
  Central foveal thickness as determined by Spectral Domain-Ocular Coherence Tomography (SD-OCT).

OTHER OUTCOMES:
Number of office visits needed | 12 months
  Number of office visits completed for patients on Arm C (treat-and-extend arm), compared to those on Arms A and B
Number of required injections | 12 months
  Number of Lucentis® injections administered to patients in Arm C, compared to those on Arms A and B

CONTACTS AND LOCATIONS:
Overall Officials: Pravin U Dugel, MD, Principal Investigator — Retinal Consultants of Arizona
Locations (4):
- United States (4):
  - Retinal Consultants of Arizona, Gilbert, Arizona
  - Retinal Consultants of Arizona, Mesa, Arizona
  - Retinal Consultants of Arizona, Peoria, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona